CLINICAL TRIAL: NCT01595477
Title: A Randomized Controlled Study of Mind-Body Skills Groups for the Treatment of War-Related Trauma in Children in Gaza
Brief Title: Mind-Body Skills Groups for the Treatment of War-Related Trauma in Children in Gaza
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Mind-Body Medicine (Other)
Collaborators: The Atlantic Philanthropies (Other)
Responsible Party: Principal Investigator, James S. Gordon, M.D., Founder and Director, The Center for Mind-Body Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC-CMBM-001
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mind-Body Skills Groups (Experimental)
  Interventions: Behavioral: Mind-Body Skills Group
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Mind-Body Skills Group — Teaching mind-body skills such as meditation, biofeedback, guided imagery, and meditation in a group setting
  Arms: Mind-Body Skills Groups

SUMMARY:
The objective of this study is to determine whether participation in a mind-body skills program by war-traumatized children in Gaza will result in improvement of posttraumatic stress symptoms, depression, and decreased hopelessness compared to a control group.

ELIGIBILITY:
Inclusion Criteria:

* having experienced a political violence or war-related criterion A stressor
* meeting the American Psychiatric Association (DSM-IV-TR) criteria for PTSD according to screening scores on the Child PTSD Symptom Scale

Exclusion Criteria:

* former psychosocial or medical treatment for mental health conditions
* significant cognitive impairment

Ages: 8 Months to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Child PTSD Symptom Scale | Change from Baseline (Week 1) at 6 weeks
Child PTSD Symptom Scale | Change from Week 6 at 18 weeks
Child PTSD Symptom Scale | Change from Baseline (Week 1) at 18 weeks

SECONDARY OUTCOMES:
Children's Depression Inventory -2 Short Form | Change from Baseline (Week 1) at 6 weeks
Children's Depression Inventory -2 Short Form | Change from Week 6 at 18 weeks
Children's Depression Inventory -2 Short Form | Change from Baseline (Week 1) at 18 weeks
Hopelessness Scale for Children | Change from Baseline (Week 1) at 6 weeks
Hopelessness Scale for Children | Change from Week 6 at 18 weeks
Hopelessness Scale for Children | Change from Baseline (Week 1) at 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James S Gordon, MD, Principal Investigator — The Center for Mind-Body Medicine
Locations (1):
- The Center for Mind-Body Medicine, Gaza City, Palestine, Israel

REFERENCES:
- See also: The Center for Mind-Body Medicine website — http://www.cmbm.org